CLINICAL TRIAL: NCT05265338
Title: A Phase I Study of KC1036 on Pharmacokinetics to Assess the Effect of High Fat Diet in Chinese Adult Healthy Subjects.
Brief Title: A Food Effect Study of KC1036 in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KC1036-I-02
Record Dates: First submitted 2022-02-16; First posted 2022-03-03 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Double cycle, self crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): In the fasting state, KC1036 po only once (60mg QD) and after 7 days，in the high fat diet state，KC1036 po only once (60mg QD).
  Interventions: Drug: KC1036
- Group B (Experimental): In the high fat diet state, KC1036 po only once (60mg QD) and after 7 days, in the fasting state, KC1036 po only once (60mg QD).
  Interventions: Drug: KC1036

INTERVENTIONS:
Drug: KC1036 — 60mg QD

SUMMARY:
The primary objective of the study was to assess the effect of High Fat Diet on the pharmacokinetics of KC1036 in Chinese adult healthy subjects.

DETAILED DESCRIPTION:
This is an open-label, randomized, two cycle self crossover experimental design study to assess the effect of High Fat Diet on the pharmacokinetics, material balance, safety of KC1036 in Chinese adult healthy subjects. This study was divided into two Groups A and B.

Group A：In the fasting state, KC1036 po only once (60mg QD) and after 7 days, in the high fat diet state, KC1036 po only once (60mg QD).

Group B：In the high fat diet state, KC1036 po only once (60mg QD) and after 7 days, in the fasting state, KC1036 po only once (60mg QD).

ELIGIBILITY:
Inclusion Criteria:

* 18~65 years of age, male.
* The weight of male subject ≥50kg, 19≤BMI≤26g/m2.
* Agree to take adequate contraceptive measures to prevent spouse pregnancy during the clinical trail.
* Able to comprehend and willing to sign an informed consent form (ICF).

Exclusion Criteria:

* Diseases such as liver, kidney, endocrine, cardiovascular, respiratory, nervous, mental, digestive tract, lung, immunity, skin, blood or metabolic disorders that are considered clinically significant by investigator, or have a history of these diseases, or have undergone major surgery, or factors that will endanger the safety of the subject or affect the research results.
* Physical examination, vital signs, laboratory examination, 12-ECG and chest film are clinically significant.
* Excessive smoking within 3 months before screening.
* History of drug and food allergy.
* Drinking 14 units of alcohol per week within 6 months prior dosing (1 unit = 360 mL of beer, or 150mL of wine).
* Participate in blood donate blood volume≥200mL or blood loss ≥200mL within 3 month prior dosing.
* Take any prescription, any over-the-counter medication, traditional Chinese medicines, vitamin products within14 days prior dosing.
* Take any clinical trial drugs within 3 months prior dosing.
* Dysphagia or history of gastrointestinal diseases affecting drug absorption.
* Combined with other viral infections (anti-HCV, anti-HIV positive, anti-TP positive, HBsAg positive) or combined with syphilis infection.
* Acute diseases requiring clinical treatment before screening or prior dosing.
* Anyone who refuse to stop ingest foods or drinks containing caffeine, alcohol from 48 hours before dosing to the end of the study.
* Urine drug positive or drug users within 3 months prior dosing.
* The investigator believes that the subjects are not eligible to participate in this trial.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 12 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) profile: Cmax | up to 13 Days
  Peak Plasma Concentration
Pharmacokinetics (PK) profile: Tmax | up to 13 Days
  Time to reach the maximum plasma concentration
Pharmacokinetics (PK) profile: T1/2 | up to 13 Days
  Terminal half-life
Pharmacokinetics (PK) profile: AUC | up to 13 Days
  Area under the single-dose plasma concentration-time curve

SECONDARY OUTCOMES:
material balance | up to 13 Days
  Drug recovery
Adverse events (AEs) | up to 43 Days
  Incidence of treatment-related AEs

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No